CLINICAL TRIAL: NCT05972304
Title: Efficiency and Safety of Nasal Positive Airway Pressure Systems During Endoscopic Procedures in High Risk Patients. Endo-Breath-Study
Brief Title: Efficiency and Safety of Nasal Positive Airway Pressure Systems During Endoscopy
Acronym: Endo-Breath
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Thomas Seufferlein, Prof. Dr. med. Benjamin Walter, University of Ulm
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EndoBreath
Record Dates: First submitted 2022-12-29; First posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Hypercapnia; Hypoxia
MeSH Terms: conditions — Hypercapnia; Hypoxia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): Patients undergoing endoscopic procedures receiving oxygen supplementation through nasal positive airway pressure system ( 10 litters/minute).
  Interventions: Device: Nasal positive airway System by Vyaire Medical
- Control Group (No Intervention): Patients undergoing endoscopic procedures receiving conventional oxygen supplementation through nasal cannula (6 litters/minute).

INTERVENTIONS:
Device: Nasal positive airway System by Vyaire Medical — Incidence of Hypercarbia and Hypoxia in interventional group and its monitoring using transcutaneous (SpO2) and (tCO2) Sensor
  Other Names: Superno2Va; Radiometer TCM 5
  Arms: Intervention Group

SUMMARY:
Goal of our study is to investigate whether the implication of nasal positive airway pressure (nPAP) system on patients with high periprocedural risk could significantly lower the incidence of severe hypoxia and hypercarbia. Furthermore, we have set up goals to assess key components and factors, which lead to development of hypercarbia during endoscopy.

DETAILED DESCRIPTION:
Sedation of high-risk patients resemble a relevant issue in interventional endoscopy.

This especially because standard oximetric monitoring displays only hypoxia and not the preceding hypercapnia. Therefore, the question arises whether the implication of a nasal positive airway pressure (nPAP) system can decrease the rate of sedation associated events.

The Null Hypothesis: The incidence of hypoxia in interventional group, using nasal positive airway pressure system, in comparison to control group with conventional oxygen supplementation canula is not significant.

Alternative Hypothesis: The incidence of hypoxia in interventional group, using nasal positive airway pressure system is significantly lower, than in a control group with conventional oxygen supplementation canula

ELIGIBILITY:
Inclusion Criteria:

* ASA III (poorly controlled Diabetes Melitus (DM) or arterial hypertension (HTN), Chronic obstructive Pulmonary Disease (COPD), morbid obesity (BMI≥40), active hepatitis, alcohol dependence or abuse, implanted pacemaker, moderate reduction of ejection fraction, End Stage Renal Disease (ESRD), Advanced Liver Disease ( ACLD) ; history (>3 months) of Myocardial Infarction, coronary artery disease (CAD) , transient ischemic attack (TIA), or CAD/stents)
* ASA IV (recent (<3 months MI, CVA, TIA, or CAD/stents, ongoing cardiac ischemia or severe valve dysfunction, severe reduction of ejection fraction, sepsis, ARD or ESRD not undergoing regularly scheduled dialysis
* Active Malignancy (ECOG Performance >2)

Exclusion Criteria:

* Patients with tracheotomy
* Pregnancy
* Intubation assisted endoscopy
* Procedure without sedation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Incidence of Hypoxia ( SpO2 < 90%, lasting longer than 10 seconds) during the endoscopic procedure | During endoscopic procedure
Incidence of severe Hypoxia ( SpO2 < 80%, lasting longer than 10 seconds) during the endoscopic procedure | During endoscopic procedure

SECONDARY OUTCOMES:
Difference of delta tcpCO2 (transcutaneous pCO2) levels between two groups | During endoscopic procedure
  Delta tcpCO2 is the difference of tpCO2 values from the beginning of the intervention to the mean tpCO2 levels observed throughout the procedure, between two groups
Number of desaturation episodes (SpO2 < 90%) | During endoscopic procedure
Interception of the intervention due to insufficient oxygenation | During endoscopic procedure
The emmergence of serious adverse events | During endoscopic procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsklinikum Ulm, Ulm, Germany

IPD SHARING:
Plan to Share IPD: No